CLINICAL TRIAL: NCT06380569
Title: A Strength-Based Intervention to Improve Job Interview Skills in Young Adults in a Community Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1139-21 Community Setting
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Gene Expression

STUDY DESIGN:
Intervention Model Description: Kessler Foundation Strength Identification and Expression (KF-STRIDE®)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): In this arm, participants would participate in in an intervention program that uses character strengths to improve job maintenance skills in young adults.
  Interventions: Behavioral: KF-STRIDE®
- Control Group (No Intervention): In this arm, participants are services as usual and will participate in their regular activities.

INTERVENTIONS:
Behavioral: KF-STRIDE® — Treatment group will receive 10 web based sessions of a strength-based training tool (once or twice a week). Sessions are approximately 60 minutes long.
  Other Names: Kessler Foundation Strength Identification and Expression
  Arms: Treatment Group

SUMMARY:
The investigators are looking to evaluate how effective a strength-based intervention may be in improving job interview skills in young adults. The investigators are examining the effects of this intervention in young adults who may have difficulty with job interviews, and who may want to improve these skills.

DETAILED DESCRIPTION:
The investigators have developed KF-STRIDE, a promising web-based intervention which focuses on helping autistic transition age youth improve interview skills by 1) learning to identify their unique employable strengths, and 2) practice speaking about those strengths to potential employers in socially appropriate ways. The inability to express one's strengths to a potential employer can negatively affect interview performance and lead to difficulty with job obtainment. Importantly, KF-STRIDE is web-based, so it is highly scalable, and uses well-established principles of positive psychology. The investigators' pilot data evaluating KF-STRIDE in a lab-based setting indicates that after using KF-STRIDE, users experience increased knowledge of their personal strengths and improved job interview skills. However, KF-STRIDE's effectiveness in a real-world setting has not been established. Kessler Foundation (KF) Center for Autism Research will partner with Spectrum Works (or other community partner) (see letter of support) to implement and evaluate KF-STRIDE in a real-world setting. Spectrum Works is a non-profit organization which provides job training and employment opportunities to autistic youth. In the current study, KF-STRIDE will be implemented at Spectrum Works (or other community partner) by Spectrum Work staff members (trained by KF staff).

ELIGIBILITY:
Inclusion Criteria:

Lives in the United States of America Between the ages of 14-26 Speaks English well and at a 4th grade reading level

Exclusion Criteria:

Had a stroke, Traumatic Brain Injury, or neurological injury or disease in the past(like brain tumor or epilepsy) Has a history of significant psychiatric illness(like schizophrenia or psychosis) Has uncontrolled seizures or other unstable medical complications

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mock Job Interview | Baseline, Immediate Post-Test between weeks 7 and 8
  Blinded reviewers using a standardized scoring measure will rate the video recorded mock job interviews
Employment Status | Baseline, Immediate Post-Test, and 6 months Post-Test
  We will examine whether the person became employed or other changes to their employment status. Yes=1, No=0
Time-to-reach Employment | 6 months Post-Test
  We will examine how long it took for the person to obtain employment. Assessed as weeks since intervention completion.
Strength Knowledge and Strengths Use Scale (SKUS) | Baseline, Immediate Post-test between weeks 7 and 8
  Measure to assess knowledge and use of one's strengths and measure changes following strengths-based interventions. Two scores: Strengths Use and Strengths Knowledge. Strengths Use values range from 14-98, with higher score indicating a better outcome. Strengths Knowledge values range from 8-56, with higher score indicating a better outcome.
Youth Interview- Self Efficacy and Anxiety | Baseline, Immediate Post-test between weeks 7 and 8
  25 items combined, about confidence and interview comfort in adolescents, with values ranging from 0 to 5 for each item, and higher scores meaning a better outcome.
Job Search Behavior Scale | Baseline, Immediate Post-test between weeks 7 and 8
  12 items measuring how often one engages in job search activities- language modified for use in youth, with values ranging from 1-5, with higher scores meaning a better outcome.
Work Readiness Scale | Baseline, Immediate Post-test between weeks 7 and 8
  13 items about the perception of one's ability to work, with values ranging from 1 to 5, with higher scores meaning a better outcome.
Global Assessment of Character Strengths (GACS) | Baseline, Immediate Post-test between weeks 7 and 8
  24 items measuring one's identification of personal character strengths, with values ranging from 1 to 5, with higher scores meaning a better outcome

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | Baseline, Immediate Post-test between weeks 7 and 8
  Self-report self-esteem questionnaire. Values range from 10-40, with higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, Ph. D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No